CLINICAL TRIAL: NCT06315101
Title: A Real-world Study of Lenvatinib Combined With Chinese Herbal Medicine for Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Effectiveness and Safety of Lenvatinib Combined With Chinese Herbal Medicine for Patients With Unresectable Hepatocellular Carcinoma: A Real-world Study in China
Status: Completed | Type: Observational
Sponsor: Guangzhou University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Donghua Liu, Director, Guangzhou University of Chinese Medicine
Other Study IDs: K-2023-092
Record Dates: First submitted 2024-03-07; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Unresectable Hepatocellular Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lenvatinib combined with Chinese Herbal Medicine
  Interventions: Drug: Chinese Herbal Medicine

INTERVENTIONS:
Drug: Chinese Herbal Medicine — Patients were treated with Chinese herbal medicine (CHM). CHM refers to the administration of a syndrome-specific herbal formula prescribed by a Traditional Chinese Medicine (TCM) physician after an uHCC diagnosis. Physicians determine the formula based on tongue and pulse examinations and personalized TCM syndromes derived from individual patient symptoms, adhering to established therapeutic principles and long-term clinical experience of physicians. The CHM formula applied in the study followed overarching TCM strategies, including reinforcing spleen qi, harmonizing liver qi, addressing blood stasis, and detoxification.

SUMMARY:
This study aims to assess the effectiveness and safety of lenvatinib plus Chinese Herbal Medicine (CHM) for patients with uHCC in China.

DETAILED DESCRIPTION:
Liver resection is one of the most important treatments for hepatocellular carcinoma (HCC). However, only a minority of patients have the opportunity to undergo surgery. The development of systemic therapy has dramatically changed the management of unresectable HCC (uHCC). And lenvatinib garners a recommendation as the primary treatment for uHCC. Many patients with uHCC in Asian countries seek complementary and alternative therapies with traditional Chinese medicine (TCM). However, the impact of lenvatinib combined with CHM on uHCC patients remains unclear. In this study, we conducted a retrospective cohort study to assess the effectiveness and safety of lenvatinib plus CHM for patients with uHCC in China.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* histologically confirmed HCC unsuitable for resection
* lenvatinib as first- or second-line therapy

Exclusion Criteria:

* patients with other primary tumors
* patients who had only one visit record and were lost to follow-up or refused follow-up
* patients with any other factors affecting study data collection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this retrospective cohort study, we collected data on consecutive patients with unresectable hepatocellular carcinoma from the electronic medical records at the First Affiliated Hospital of Guangzhou University of Chinese Medicine in China, covering the period from September 2018 to July 2022, and conducted follow-ups until May 30, 2023. All cases underwent lenvatinib combined with CHM as first-line therapy, with or without PD-1 inhibitors.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy outcomes | after 8 weeks of the initiation of Lenvatinib combined with Chinese Herbal Medicine
  Tumor Response after 8 weeks of treatment according to the modified Response Evaluation Criteria in Solid Tumor (mRECIST)
Survival analysis | 2022/10/01-2023/12/31
  Kaplan-Meier estimates of overall survival (OS)
Survival analysis | 2022/10/01-2023/12/31
  Kaplan-Meier estimates of progression-free survival (PFS)

SECONDARY OUTCOMES:
Adverse Events assessment | after 8 weeks of the initiation of Lenvatinib combined with Chinese Herbal Medicine
  Adverse Events (AEs) were assessed following the guidelines of the Common Terminology Criteria for Adverse Events version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Suihui Li, postgraduate, Study Director — The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine
Locations (1):
- the First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No